CLINICAL TRIAL: NCT05710848
Title: A Phase 1/2a Study of STM-416 Administered Intraoperatively to Patients Undergoing Transurethral Resection of Bladder Tumor (TURBT) for Recurrent High-Grade Papillary Bladder Cancer
Brief Title: A Study of STM-416 Administered to Patients Undergoing TURBT for Recurrent Bladder Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SURGE Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STM-416-01
Record Dates: First submitted 2022-12-15; First posted 2023-02-02 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-07

CONDITIONS: Non-muscle-invasive Bladder Cancer
Keywords: Open-label; Dose escalation; STM-416; Resiquimod; Toll-like receptor 7/8; Non-Muscle Invasive Bladder Cancer; TURBT; Immunotherapy; BCG
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Singe group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- STM-416 (Experimental): STM-416
  Interventions: Drug: STM-416

INTERVENTIONS:
Drug: STM-416 — STM-416 monotherapy

SUMMARY:
This is a first-in-human (FIH), Phase 1/2a, multi center, open-label, single treatment, dose escalation and expansion study designed to determine the safety and tolerability of STM-416 in patients with bladder cancer.

DETAILED DESCRIPTION:
This is a 2-part, multicenter, first-in-human (FIH), Phase 1/2a study in patients with a history of pathologically confirmed high-grade Ta or T1 NMIBC without CIS who have completed SOC previously, with recurrent papillary disease seen on cystoscopy, and who are undergoing TURBT without perioperative intravesical chemotherapy. All patients will receive relevant SOC therapy following TURBT. SOC will be administered in the adjuvant setting.

Phase 1 is an open-label, single-treatment, dose-escalation study to evaluate the safety and tolerability of up to 6 increasing doses of intraoperatively administered STM-416 utilizing a 3+3 convention, with 3 to 6 patients enrolled in each STM-416 dose level, with a minimum of 6 patients enrolled at the highest dose level, for a total of approximately 30 patients.

Phase 2a is a randomized, single-blind, single-treatment, dose-expansion study that will comprise 2 arms: TURBT + STM-416 Dose 1 followed by SOC versus TURBT + STM-416 Dose 2 followed by SOC.

ELIGIBILITY:
Inclusion Criteria:

1. Are aged 18 years or older;
2. Have a history of pathologically confirmed high-grade Ta or T1 NMIBC without CIS who have completed SOC previously, with recurrent papillary disease seen on cystoscopy, and who are undergoing TURBT without perioperative intravesical chemotherapy;
3. Are considered high risk for recurrence;
4. Have Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2;
5. Have adequate organ and marrow function as defined below:

   * Hemoglobin 9.0 g/dL;
   * Absolute neutrophil count 1.5 × 109/L (1500 per mm3);
   * Platelet count 75 × 109/L (75,000 per mm3);
   * Serum bilirubin 1.5 × institutional upper limit of normal (ULN);
   * AST (serum glutamic-oxaloacetic transaminase)/ALT (serum glutamic-pyruvic transaminase) 2.5 × institutional ULN; and
   * Creatinine CL 60 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine CL: Males: Creatinine CL (mL/min) = Weight (kg) × (140 - Age)/72 × serum creatinine (mg/dL); or Females: Creatinine CL (mL/min) = Weight (kg) × (140 - Age) × 0.85/72 × serum creatinine (mg/dL).

Exclusion Criteria:

1. Have a history of CIS or MIBC;
2. Are receiving any other investigational agents;
3. Have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to resiquimod (R848), or excipients used in STM-416 including poloxamer 407 and sodium hyaluronate;
4. Have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

   Urinary tract infections are not exclusionary unless they are NCI-CTCAE Grade 3 or higher;
5. Are a woman of childbearing potential regardless of contraceptive use; Note: Women of childbearing potential are only to be excluded in Phase 1 and Phase 2a to avoid bias due to the low prevalence of NMIBC in this population. However, they will be included in subsequent Phase 2/3 studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women of childbearing potential are only to be excluded in Phase 1 and Phase 2a to avoid bias due to the low prevalence of NMIBC in this population.
Enrollment: 75 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) [Safety and Tolerability] Phase 1 | 21 days
  Incidence of dose-limiting toxicities (DLTs) over the first 21-days of study treatment
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] Phase 1 | Time on trial up to 90 days
  Incidence of serious adverse events (SAEs), and adverse events (AEs), graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0
Recurrence free survival time (Phase 2a) | Through study completion up to 24 months
  Recurrence will be evaluated by cystoscopy and urine cytology

SECONDARY OUTCOMES:
Pharmacokinetics of STM-416 (Phase 1) | Day 0, post 24 hours, post 48 hour
  Maximum plasma concentration (Cmax) of resiquimod (R848) in patient blood for the single dose level (Phase 1)
Pharmacokinetics of STM-416 (Phase 1) | Day 0, post 24 hours, post 24 hour
  Area under the plasma concentration versus time curve (AUC) of resiquimod (R848) in patient blood for the single dose level (Phase 1)
Pharmacodynamics of STM-416 | Day 0, post 24 hours, post 48 hours, post 21 days, post 90 days
  Pharmacodynamic assessments in plasma and urine will be listed and summarized by dose level for Phase 1/2a

CONTACTS AND LOCATIONS:
Overall Officials: Seth Lerner, MD, Principal Investigator — Baylor College of Medicine
Locations (10):
- United States (10):
  - Arizona Urology Specialists, Tucson, Arizona
  - University of Florida, Gainesville, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Duke Cancer Center, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates, P.C., Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist, Houston, Texas

IPD SHARING:
Plan to Share IPD: No